CLINICAL TRIAL: NCT04376307
Title: The Effects of Minimal Flow Anesthesia on Hemodynamic Parameters, Compilation and Gas Consumption in Single Lung Ventilation
Brief Title: Minimal Flow Application in One Lung Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Fatih Dogu Geyik, MD, Principal Investigator, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/514/172/15
Record Dates: First submitted 2020-04-24; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Ventilator Lung; Anesthesia; Functional
Keywords: one lung ventilation; low flow anesthesia; gas consumption

STUDY DESIGN:
Intervention Model Description: prospectice randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- minimal flow anesthesia (Experimental): the patiennts who have thoracic sugery with one lung ventilaiton
  Interventions: Procedure: minimal flow anesthesia

INTERVENTIONS:
Procedure: minimal flow anesthesia — Investigators will use minimal flow anesthesia (0,5 lt/min) during surgery with one lung ventilation

SUMMARY:
Interest in low fresh gas flow anesthesia has increased in recent years. The high standard of anesthesia machines, the presence of monitors that continuously and thoroughly analyze the anesthetic gas composition, and the increased knowledge of the pharmacodynamics and pharmacokinetics of inhalation anesthetics greatly facilitated the safe administration of low-flow anesthesia.Low-flow anesthesia can be mentioned for most patients if modern re-breathing systems are used but only if the fresh gas flow rate is reduced below 2 lt / min. In 1974, Virtue was defined as a technique called minimal flow, in which the fresh gas flow was not exceeded 0.5 lt / min. Although there are too many applications for low current in the literature, there is little literature for use in one lung.

DETAILED DESCRIPTION:
Our research is planned prospectively. During the preoperative examination, patients will be informed about the study and their written consent will be obtained. On the morning of the operation, anesthesia gas monitor calibration and leak test will be started with automatic tests of the anesthesia device (Drager-Perseus A500).The leak test for the ventilator and breathing circuit for the patient will be repeated in all operations. The carbon dioxide trap will be evaluated in terms of its dryness and color and will be replaced at appropriate times. The patients who were taken to the operation table were venously opened with a 20-gauge cannula from the back of the hand, and perfusion of 10 ml / kg / h 0.9% sodium chloride was started. ECG, SPO2, NIBP monitoring (Siemens SC-7700), starting before anesthesia (basal), after induction, after intubation 1.min and 5., 10., 15., 20., 25., 30., 40 ., 50th, 60th, 75th, 90th, 105th, 120th minutes and preoperative arterial blood gas (AKG) will be taken.1μg / kg fentanyl (Fentanyl Citrate, Abbott Lab. North Chicago, USA), 5-7 mg / kg thiopental (Pental) for anesthesia induction after preoxygenation in 100% O2 and fresh gas flow 4L / min with spontaneous breathing for 3 minutes with mask sodium, IE Ulagay, Istanbul, Turkey) and 0.1 mg / kg vecuronium (Norcuro, Organon, Oss. the Netherlands) was administered iv. When muscle relaxation was observed, orotracheal intubation was performed and the patient (Dräger Perseus) was adjusted with an anesthesia device to have a tidal volume of 7-10 ml / kg, respiratory frequency 12 / min, and the ratio of I: E 1: 2. The tube was placed by selective intubation with the help of fiberoptic bronchoscopy. MAC values will be kept between 4-6%. Alarm limits FiO2 30% lower limit, desflurane 10% vol upper limit, EtCO2 45mmhg upper limit Paw 5cmh20 six lower limit, 30cmh2o upper limit set. co2 absorbent, as sodalime (Sorbo-lime, Berk, Turkey) were used.

Arterial Blood Gas (ABG) analysis will be performed at zero and then half hour intervals of single lung ventilation. Special attention will be paid not to open the system. Muscle relaxant antagonism will be achieved in all patients with 0.01mg / kg of atropine and 0.03mg / kg of neostigmine. At the end of the operation, the recovery period characteristics of all patients at the 1st, 5th, and 10th minutes before and after extubation were evaluated with Aldrete Kraulik's post-anesthesia evaluation system. Gas consumption amounts will be monitored on the monitor and recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3 Patients
* Single lung ventilation during the operation
* Age>18

Exclusion Criteria:

Age<18

* ASA 4
* pregnancy
* COPD patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Age | during surgery
  Years
Gender | during surgery
  Male/Female
ASA : | during surgery
  I, II, III, IV
Height: | during surgery
  centimeter
Weight | during surgery
  kilogram
BMI: | during surgery
  kg/m2
Side of surgery | during surgery
  left /right
Side of double lumen tube | during surgery
  left/right
Desfluran consumption | during surgery
  ml
Heart Rate | during surgery
  beats /minute
SpO2 | during surgery
  percent
Systolic Blood Pressure | during surgery
  mmHg/min
Diastolic Blood Pressure | during surgery
  mmHg/min
Respiratory Rate | during surgery
  frequency/ min
Intubation tube size | during surgery
  french
duration of anesthesia | during surgery
  minutes
Duration of single lung ventilation | during surgery
  minutes
Operation time | during surgery
  minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Kartal Dr. Lutfi Kirdar Education and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Baum JA. Low-flow anesthesia: theory, practice, technical preconditions, advantages, and foreign gas accumulation. J Anesth. 1999;13(3):166-74. doi: 10.1007/s005400050050. No abstract available. PMID 14530937
- [Background] Honemann CW, Hahnenkamp K, Mollhoff T, Baum JA. Minimal-flow anaesthesia with controlled ventilation: comparison between laryngeal mask airway and endotracheal tube. Eur J Anaesthesiol. 2001 Jul;18(7):458-66. doi: 10.1046/j.1365-2346.2001.00868.x. PMID 11437874